CLINICAL TRIAL: NCT00012805
Title: Effectiveness and Cost Impact of a Telecommunications System in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: IIR 97-022
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Lung Diseases, Obstructive
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Telephone Monitoring

INTERVENTIONS:
Procedure: Telephone Monitoring

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the most common chronic illnesses among veterans in the adult population, and accounts for substantial morbidity and mortality in this population. Interventions that enhance symptom self-monitoring and increase understanding of COPD therapy may lead to earlier detection of clinical deterioration permitting more timely intervention by health care providers. However, such interventions are labor-intensive and expensive, and typically require patients to go to a medical facility on a regular basis. A novel means of providing such interventions is a Telephone-Linked Computer (TLC) system, a computer-based telecommunications system that can monitor, educate, and counsel patients through regular automated conversations in patients� homes. In previous studies, we have demonstrated the applicability of TLC technology in the clinical monitoring of adults with chronic disease conditions such as hypertension and hypercholesterolemia.

DETAILED DESCRIPTION:
Background:

Chronic obstructive pulmonary disease (COPD) is one of the most common chronic illnesses among veterans in the adult population, and accounts for substantial morbidity and mortality in this population. Interventions that enhance symptom self-monitoring and increase understanding of COPD therapy may lead to earlier detection of clinical deterioration permitting more timely intervention by health care providers. However, such interventions are labor-intensive and expensive, and typically require patients to go to a medical facility on a regular basis. A novel means of providing such interventions is a Telephone-Linked Computer (TLC) system, a computer-based telecommunications system that can monitor, educate, and counsel patients through regular automated conversations in patients� homes. In previous studies, we have demonstrated the applicability of TLC technology in the clinical monitoring of adults with chronic disease conditions such as hypertension and hypercholesterolemia.

Objectives:

The objectives of the study were to determine whether a telecommunications system for COPD care (TLC-COPD) leads to improvements in functional status and quality of life (QOL) as well as to reductions in health care utilization and costs exceeding the TLC intervention.

Methods:

The study was designed in the form of a randomized controlled trial involving subjects with COPD who receive care at two Boston-area VA hospitals. Subjects were assigned to either TLC-COPD or a usual care control group.

Status:

Complete.

ELIGIBILITY:
Inclusion Criteria:

COPD diagnosis; FEV, < _65% pred; FEV, /FVC<_85% pred

Exclusion Criteria:

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David William Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States